CLINICAL TRIAL: NCT02889055
Title: Evaluation of Mirus™ for Sedation in Resuscitation
Acronym: MIRUS
Status: Terminated | Type: Observational
Why Stopped: Safety profile was not satisfying with sevolflurane
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC15.111
Record Dates: First submitted 2016-08-03; First posted 2016-09-05 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Patient Requiring Mechanical Ventilation
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: patient requiring the MIRUS (mechanical ventilation)

SUMMARY:
Current recommendations for the conduct of sédationanalgésie ICU encourage the use of the lightest possible sedation strategies, avoiding the administration of benzodiazepines source of longer durations of ventilation and ICU stay of syndrome cessation, mental confusion. Among the proposed alternatives, administration of halogenated volatile agents (sevoflurane) in resuscitation is interesting because their favorable pharmacokinetic even after prolonged administration: no tachyphylaxis, rapid clearance, no withdrawal syndrome.

There are two suitable delivery devices sevoflurane in intensive care, both with CE marking. The device Mirus ™ (Pall Medical, Fribourg, Switzerland) is the newest and it is easy to use and reliable. The objective of this study was to evaluate the use of Mirus ™ device in trauma resuscitation and cardiovascular resuscitation.

Specifically, it will use this modality in case of failure with conventional sedation products (propofol, midazolam): maximum permissible doses, sedation weaning failure due to severe agitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* In mechanical ventilation for more than 48 hours
* No intracranial hypertension
* In severe state of agitation measured by a sedation scale score greater than 2 RASS
* Agitation observed in two circumstances: receiving maximal doses of propofol (≥ 5 mg / kg / h) and / or midazolam (≥ 0.2 mg / kg / h), or weaning failure to stop the sedation agitation.

Exclusion Criteria:

* Presence of a severe head injury (Glasgow initial score between 3 and 8) requiring monitoring intracranial pressure and / or treatment of intracranial hypertension
* Sedation with dexmedetomidine
* Personal or family antecedent of anesthetic malignant hyperthermia
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient requiring mechanical ventilation for more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-01-17 (Actual); Primary Completion 2016-10-08 (Actual); Study Completion 2016-10-08 (Actual)

PRIMARY OUTCOMES:
ead-time (in minutes) of sevoflurane sedation for obtaining a target RASS score between 1 (anxious) and 2 (mild sedation). | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François PAYEN, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Kong KL, Willatts SM, Prys-Roberts C. Isoflurane compared with midazolam for sedation in the intensive care unit. BMJ. 1989 May 13;298(6683):1277-80. doi: 10.1136/bmj.298.6683.1277. PMID 2500195
- [Background] Sackey PV, Martling CR, Carlsward C, Sundin O, Radell PJ. Short- and long-term follow-up of intensive care unit patients after sedation with isoflurane and midazolam--a pilot study. Crit Care Med. 2008 Mar;36(3):801-6. doi: 10.1097/CCM.0B013E3181652FEE. PMID 18431266
- [Background] Sackey PV, Martling CR, Granath F, Radell PJ. Prolonged isoflurane sedation of intensive care unit patients with the Anesthetic Conserving Device. Crit Care Med. 2004 Nov;32(11):2241-6. doi: 10.1097/01.ccm.0000145951.76082.77. PMID 15640636
- [Background] Mesnil M, Capdevila X, Bringuier S, Trine PO, Falquet Y, Charbit J, Roustan JP, Chanques G, Jaber S. Long-term sedation in intensive care unit: a randomized comparison between inhaled sevoflurane and intravenous propofol or midazolam. Intensive Care Med. 2011 Jun;37(6):933-41. doi: 10.1007/s00134-011-2187-3. Epub 2011 Mar 29. PMID 21445642
- [Background] Rohm KD, Wolf MW, Schollhorn T, Schellhaass A, Boldt J, Piper SN. Short-term sevoflurane sedation using the Anaesthetic Conserving Device after cardiothoracic surgery. Intensive Care Med. 2008 Sep;34(9):1683-9. doi: 10.1007/s00134-008-1157-x. Epub 2008 May 24. PMID 18500419
- [Background] Hellstrom J, Owall A, Bergstrom J, Sackey PV. Cardiac outcome after sevoflurane versus propofol sedation following coronary bypass surgery: a pilot study. Acta Anaesthesiol Scand. 2011 Apr;55(4):460-7. doi: 10.1111/j.1399-6576.2011.02405.x. Epub 2011 Feb 22. PMID 21342154
- [Background] Soukup J, Scharff K, Kubosch K, Pohl C, Bomplitz M, Kompardt J. State of the art: sedation concepts with volatile anesthetics in critically Ill patients. J Crit Care. 2009 Dec;24(4):535-44. doi: 10.1016/j.jcrc.2009.01.003. Epub 2009 Mar 27. PMID 19327951
- [Background] Perbet S, Bourdeaux D, Sautou V, Pereira B, Chabanne R, Constantin JM, Chopineau J, Bazin JE. A pharmacokinetic study of 48-hour sevoflurane inhalation using a disposable delivery system (AnaConDa(R)) in ICU patients. Minerva Anestesiol. 2014 Jun;80(6):655-65. Epub 2013 Nov 13. PMID 24226486
- [Background] Chabanne R, Perbet S, Futier E, Ben Said NA, Jaber S, Bazin JE, Pereira B, Constantin JM. Impact of the anesthetic conserving device on respiratory parameters and work of breathing in critically ill patients under light sedation with sevoflurane. Anesthesiology. 2014 Oct;121(4):808-16. doi: 10.1097/ALN.0000000000000394. PMID 25111218
- [Background] Sackey PV, Martling CR, Nise G, Radell PJ. Ambient isoflurane pollution and isoflurane consumption during intensive care unit sedation with the Anesthetic Conserving Device. Crit Care Med. 2005 Mar;33(3):585-90. doi: 10.1097/01.ccm.0000156294.92415.e2. PMID 15753751
- [Background] Berton J, Sargentini C, Nguyen JL, Belii A, Beydon L. AnaConDa reflection filter: bench and patient evaluation of safety and volatile anesthetic conservation. Anesth Analg. 2007 Jan;104(1):130-4. doi: 10.1213/01.ane.0000248221.44383.43. PMID 17179257
- [Background] Bomberg H, Glas M, Groesdonk VH, Bellgardt M, Schwarz J, Volk T, Meiser A. A novel device for target controlled administration and reflection of desflurane--the Mirus. Anaesthesia. 2014 Nov;69(11):1241-50. doi: 10.1111/anae.12798. Epub 2014 Jul 9. PMID 25040673